CLINICAL TRIAL: NCT04655534
Title: The Effect of Inspiratory Muscle Warm-Up Prior to Inspiratory Muscle Training in Addition to Exercise Training in Patients With COPD
Brief Title: The Effect of Inspiratory Muscle Warm-Up in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Ridvan Aktan, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RidvanAKTAN_2018.KB.SAG.026
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD
Keywords: inspiratory muscle warm-up; inspiratory muscle training; lung functions; respiratory functions; respiratory muscle strength; exercise capacity; dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Intervention Model Description: This study was designed as a prospective and experimental study. Participants were randomly divided into two groups as the study group (IMW Group) and the control group (Standard IMT Group). The Standard IMT Group performed only inspiratory muscle training (IMT), while the IMW Group performed an inspiratory muscle warm-up (IMW) protocol for warming the inspiratory muscles before each IMT session. The IMT and IMW applied using a threshold pressure loading device.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMW Group (Experimental): Patients who performed inspiratory muscle warm-up (IMW) before inspiratory muscle training (IMT)
  Interventions: Other: Inspiratory Muscle Warm-up (IMW); Other: Inspiratory Muscle Training (IMT); Other: Respiratory exercises and aerobic exercise program
- Standart IMT Group (Experimental): Patients who performed standard inspiratory muscle training (IMT) without inspiratory muscle warm-up (IMW) protocol
  Interventions: Other: Inspiratory Muscle Training (IMT); Other: Respiratory exercises and aerobic exercise program

INTERVENTIONS:
Other: Inspiratory Muscle Warm-up (IMW) — The IMW protocol applied before each inspiratory muscle training (IMT) session by using a threshold inspiratory muscle trainer. The IMW protocol consists of 2 sets of 30 breaths in 40% of the maximal inspiratory pressure (MIP), with 1 min rest between sets. The intensity of MIP adjusted by two weekly MIP measurements.
  Arms: IMW Group
Other: Inspiratory Muscle Training (IMT) — The IMT applied twice a day as 30 breath repetitions at 60% of the maximal inspiratory pressure (MIP). The intensity of MIP adjusted by two weekly MIP measurements.
Other: Respiratory exercises and aerobic exercise program — Then the respiratory exercises and aerobic exercise program performed in both groups in each session. Aerobic exercise program; After 5 min of general body warming, applied 20 min with a load of 4-6 according to the modified Borg scale on the treadmill, finished with 5 min whole body cool-down. All program applied to 3 days a week for 8 weeks under the supervision of a physiotherapist and other days of the week without a supervisor.

SUMMARY:
In this study, it is aimed to investigate the effect of inspiratory muscle warm-up (IMW) performed before inspiratory muscle training (IMT) in addition to general exercise training on respiratory functions, respiratory muscle strength, exercise capacity, perceived dyspnea intensity and health-related quality of life in patients with COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a disease that leads to increased morbidity and mortality with severe pulmonary complications. The Global Burden of Disease studies have estimated that COPD is the third leading cause of death worldwide. The effects of COPD are not only limited to the lungs but also affects other organs and systems, causing loss of strength in the respiratory and peripheral muscles, which leading to a decreased capacity for exercise. Respiratory muscles are the skeletal muscles that can be trained based on the principles of exercise just like peripheral muscles. It is known that while doing exercise training in peripheral muscles, more muscle performance can be achieved by warming up those muscles before the loading phase. In this study, it is aimed to investigate the effect of inspiratory muscle warm-up (IMW) performed before inspiratory muscle training (IMT) in addition to general exercise training on respiratory functions, respiratory muscle strength, exercise capacity, perceived dyspnea intensity and health-related quality of life in patients with COPD.

Participants were randomly divided into two groups as the study group (IMW Group) and the control group (Standard IMT Group). The Standard IMT Group performed only IMT, while the IMW Group performed an IMW protocol for warming the inspiratory muscles before each IMT session. The IMT and IMW were applied using a threshold pressure loading device. The IMT applied as 30 breath repetitions at 60% of the maximal inspiratory pressure (MIP). The intensity of MIP adjusts by two weekly MIP measurements. The protocol of IMW consists of 2 sets of 30 breaths at 40% of MIP, with 1 min rest between sets, using a threshold inspiratory muscle trainer. Then the respiratory exercises and aerobic exercise program performed in both groups in each session. Aerobic exercise program; After 5 min of general body warming, applied 20 min with a load of 4-6 according to the modified Borg scale on the treadmill, finished with 5 min whole body cool-down. All program applied to 3 days a week for 8 weeks under the supervision of a physiotherapist and other days of the week without a supervisor. Demographic features questioned and recorded in the data recording form through a mutual interview in patients who meet the inclusion criteria. All patients evaluated before treatment and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosing COPD in accordance with Global initiative for chronic obstructive pulmonary disease (GOLD) guideline criteria
* Having a Maximal inspiratory pressure (MIP) less than 60 cmH2O
* Aged between 45 and 70 years
* Independent mobilization
* Volunteering to research
* Stable clinical condition (same medication routine without taking any antibiotics for the last 3 weeks and/or no acute exacerbation in the last 3 months)

Exclusion Criteria:

* Not quitting smoking
* A previous pneumonectomy or lobectomy operation.
* Pneumonia in the last 3 months.
* Any pulmonary infection during the study.
* Requirement for supplemental oxygen therapy
* Orthopaedic or neurological conditions effecting the ability to exercise

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
Respiratory functions | 8 weeks
  Respiratory functions were evaluated by pulmonary function tests. Pulmonary function tests were performed in accordance with the American Thoracic Society (ATS) / European Respiratory Society (ERS) criteria, in a sitting position with a computer-compatible spirometer (Sensor Medics Vmax 22 machine, SensorMedics Inc., Anaheim, CA). Percentages of forced expiratory volume in one second (FEV1), forced vital capacity (FVC) and FEV1 / FVC ratio values relative to the predicted value were recorded in pulmonary function tests.
Inspiratory muscle strength | 8 weeks
  Inspiratory muscle strength (MIP) was measured using a hand-held mouth pressure device (Micro RMP; Micro Medical, Rochester, UK). Three to five acceptable and reproducible maximal manoeuvres (i.e., differences between values <10%) were performed and the highest value was recorded.
Expiratory muscle strength | 8 weeks
  Expiratory muscle strength (MEP) was measured using a hand-held mouth pressure device (Micro RMP; Micro Medical, Rochester, UK). Three to five acceptable and reproducible maximal manoeuvres (i.e., differences between values <10%) were performed and the highest value was recorded.
Dyspnea assessment | 8 weeks
  The modified Medical Research Council (mMRC) Dyspnea Scale was used to evaluate the severity of dyspnea. Commonly used in the assessment of dyspnea in COPD, mMRC has a five-level scoring system ranging from 0 to 4. A high score indicates an increased sense of dyspnea.
Exercise capacity assessment | 8 weeks
  The 6-Minute Walking Test distance (6MWD) was used to assess exercise capacity.

SECONDARY OUTCOMES:
Health-Related Quality of Life (HRQOL) using the 36-item Short Form Survey (SF-36) | 8 weeks
  The SF-36 is a general quality of life survey which includes 36 items and enables the measurement of eight sections; physical functioning, social role functioning, physical role functioning, emotional role functioning, mental health, vitality, bodily pain and general health perceptions. Each category is scored from 0 to 100. Lower scores indicating worse HRQOL.
Health-Related Quality of Life assessment using the St. George's Respiratory Questionnaire (SGRQ) | 8 weeks
  The SGRQ is a specific questionnaire for respiratory diseases. It is a self-administered questionnaire by patients which questioned 50 items with 76 weighted responses divided into three areas: symptoms (8 items), activities (16 items), effects of the disease (26 items). The three parts of the questionnaire are scored separately and the total score is calculated. Scores range from 0-100. Higher scores indicating worse HRQOL.

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Ozalevli, PT, Prof, Study Director — Dokuz Eylul University; Ridvan Aktan, PT, PhD, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bisca GW, Camillo CA, Cavalheri V, Pitta F, Osadnik CR. Peripheral muscle training in patients with chronic obstructive pulmonary disease: novel approaches and recent advances. Expert Rev Respir Med. 2017 May;11(5):413-423. doi: 10.1080/17476348.2017.1317598. Epub 2017 Apr 17. PMID 28385046
- [Background] Volianitis S, McConnell AK, Koutedakis Y, Jones DA. Specific respiratory warm-up improves rowing performance and exertional dyspnea. Med Sci Sports Exerc. 2001 Jul;33(7):1189-93. doi: 10.1097/00005768-200107000-00017. PMID 11445767
- [Background] Ross EZ, Nowicky AV, McConnell AK. Influence of acute inspiratory loading upon diaphragm motor-evoked potentials in healthy humans. J Appl Physiol (1985). 2007 May;102(5):1883-90. doi: 10.1152/japplphysiol.00694.2006. Epub 2007 Jan 18. PMID 17234806
- [Background] Ozdal M. Acute effects of inspiratory muscle warm-up on pulmonary function in healthy subjects. Respir Physiol Neurobiol. 2016 Jun 15;227:23-6. doi: 10.1016/j.resp.2016.02.006. Epub 2016 Feb 21. PMID 26903486
- [Background] Volianitis S, McConnell AK, Jones DA. Assessment of maximum inspiratory pressure. Prior submaximal respiratory muscle activity ('warm-up') enhances maximum inspiratory activity and attenuates the learning effect of repeated measurement. Respiration. 2001;68(1):22-7. doi: 10.1159/000050458. PMID 11223726
- [Background] Lomax M, Grant I, Corbett J. Inspiratory muscle warm-up and inspiratory muscle training: separate and combined effects on intermittent running to exhaustion. J Sports Sci. 2011 Mar;29(6):563-9. doi: 10.1080/02640414.2010.543911. PMID 21347970